CLINICAL TRIAL: NCT06648408
Title: Effects of Ballet Training on Kinematics and Subjective Parameters in Children With Idiopathic Coxa Antetorta: a Randomized Controlled Trial
Brief Title: Ballet Training in Children With Idiopathic Coxa Antetorta
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00689; ks24Widmer
Record Dates: First submitted 2024-10-14; First posted 2024-10-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Femoral Anteversion
Keywords: Increased femoral anteversion (IFA); Idiopathic coxa antetorta; Childhood knee pain; Physical activity intervention; Ballet training for children; Hip strength and mobility; Knee flexion in children; Exercise for hip flexibility; In-toeing gait in children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ballet training (Experimental): The children in this arm of the study will receive ballet training.
  Interventions: Procedure: Balett Training
- Control group (No Intervention): The children in the control group in this study will not receive any intervention, according to the German guidelines for idiopathic coxa antetorta 2002. This is in line with the standard approach, as children in this developmental phase typically do not receive therapy for this condition.

INTERVENTIONS:
Procedure: Balett Training — The ballet training will happen twice a week for six weeks, with each session lasting 60 minutes, for a total of 12 sessions. These sessions will be held in groups of 10 to 12 children and led by experienced ballet teachers. The classes will follow a beginner-level ballet routine, introducing the kids to ballet techniques in a fun and playful way, making sure they learn the movements step by step. Each lesson will follow the same structure, allowing the children to improve their skills week after week. In addition to the group sessions, the children will be given a 10-minute daily home exercise program. This will include simple ballet exercises they learned in their first class, which they should practice on the five days when they don't have ballet sessions. The children will track their practice in a child-friendly diary designed just for them.
  Arms: Ballet training

SUMMARY:
This study looks at how ballet training affects movement and personal feelings in children with a condition called idiopathic coxa antetorta.

DETAILED DESCRIPTION:
Increased femoral anteversion (IFA) occurs when the top of the thigh bone tilts forward more than normal. Many healthy kids and teens aren't considered to have a problem with this as long as they show no symptoms, since it often corrects itself by the time they reach ages 12 to 14. However, experts believe this condition might lead to complications later in life. Research indicates that children with IFA may be more prone to issues like kneecap misalignment, knee pain, and even arthritis as they grow older. This is likely due to the way their knees bend differently when they walk. Kids with IFA often walk with their toes pointing inward, which increases their chances of tripping and falling. They may also experience pain that interferes with their daily activities. It is assumed that strengthening the hips and improving hip flexibility could help reduce the need for compensatory movements, ultimately lowering the risk of tripping, falling, and experiencing pain in everyday life. This study is a randomized controlled trial aimed at examining how ballet training influences knee movement-specifically knee flexion-during walking in children with idiopathic coxa antetorta. The goal is to determine whether ballet training enhances the children's overall mobility and how they feel about their ability to move. Additionally, the study seeks to find out how this training can be effectively incorporated into the daily routines of affected schoolchildren.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic coxa antetorta with FNA> 30°
* Children between 8 and 12 years of age
* Cognitive abilities must include: Ability to actively participate in a 60-minute ballet class; Ability to communicate pain or discomfort; Ability to attend training, testing and follow-up sessions. All included participants can make decisions on their own and do not show any signs of mental or cognitive limitations.

Exclusion Criteria:

* Any surgery within 6 months prior to the start of the study or surgery scheduled during the study period. Other medications can be continued as prescribed by the participants' physician
* Known cardiovascular or pulmonary diseases that have not received medical clearance to participate in the physical exercise intervention
* Neurological or other musculoskeletal comorbidities
* The children should not have completed any ballet training in the last 12 months
* Pregnancy

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Kinematic measurement and | Week1 and week 8
  This study will track knee flexion during the mid-stance phase of walking, as children with coxa antetorta often show increased knee bending, which can lead to future knee issues. The children's walking will be recorded using a 2D gait analysis system on the C-Mill treadmill, offering accurate results while minimizing stress and reducing the chance of errors.
Subjective functional mobility | Week1 and week 8
  The children's mobility and quality of life will be assessed, using the parent-reported Pediatric Outcomes Data Collection Instrument (PODCI), a reliable questionnaire designed for children with musculoskeletal conditions. It measures various aspects of daily functioning and well-being, and the scores range from 0 to 100, with lower scores indicating more difficulties.

SECONDARY OUTCOMES:
Gait Analysis | Week1 and week 8
  Gait analysis will be performed on the C-Mill by Motek treadmill. To ensure safety while determining the speed at which a stumble might occur, the children will be secured with a harness to prevent falls or injuries.
Measurement of femoral anteversion angle (°) | Week1 and week 8
  The femoral neck anteversion (FNA) will be measured using Craig's test, where we assess the angle at the prominent part of the hip while the child lies face down with their knee bent.
Measurement of hip strength (N) | Week1 and week 8
  The maximum strength of the hip flexors, extensors, external rotators, and abductors will be measured using dynamometers, which are reliable tools for checking how strong these muscles are.
Measurement of hip mobility (°) | Week1 and week 8
  The passive range of motion for internal and external rotation will be measured using a goniometer while the participants lie face down with their hip straight and knee bent at a 90° angle.
Feasibility assessment | Week 8
  To evaluate how feasible the intervention is, the number of training sessions the children actually attend will be tracked and compared to the planned sessions and calculate the attendance rate. The ballet teacher will maintain an attendance list, and the children will also record their participation in a specially designed, child-friendly diary.

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Widmer, Dr. med., Principal Investigator — Universitäts-Kinderspital beider Basel (UKBB)
Locations (1):
- Universitäts-Kinderspital beider Basel (UKBB), Basel, Switzerland